CLINICAL TRIAL: NCT02662972
Title: Botulinum Toxin Type A Block of the Sphenopalatine Ganglion in Trigeminal Neuralgia. Safety Issues.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTATN2015; 2015-002643-33 (EudraCT Number)
Record Dates: First submitted 2015-11-26; First posted 2016-01-26 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Trigeminal Neuralgia; Headache Disorders
Keywords: Nerve block; Sphenopalatine Ganglion Block; Botulinum Toxins, Type A
MeSH Terms: conditions — Trigeminal Neuralgia; Headache Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Botulinum Toxin (Experimental): The patients will be injected with 25 IU of Botulinum Toxin Type A towards the sphenopalatine ganglion in the affected side (ipsilateral to the pain)
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A
  Other Names: Botox; BTA

SUMMARY:
Trigeminal neuralgia is one of the strongest pains known to humans. Some patients do not have enough effect with the available pharmaceutical treatments and are offered surgery. There are different types of procedures and most of them are complex with a risk for complications. The researchers want to start a pilot study on 10 patients with a new surgical technique using neuronavigation. The target will be a neural structure (sphenopalatine ganglion) which has an important role in facial pain. There have been a few trials trying to block this structure in trigeminal neuralgia, but none using this new approach with botulinum toxin. The researchers technique requires local anesthesia only (awake patient). The researchers believe that this treatment can become a "low threshold"-treatment for patients who do not have enough effect with pharmacological treatment and a better alternative to other complex surgical approaches. Using this new neuronavigation system the researchers can reach this neural structure with high precision.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent
* Trigeminal neuralgia defined in International Classification of Headache Disorders (ICHD)-3 criteria
* Unsatisfactory effect of pharmacological treatment

Exclusion Criteria:

* Microvascular decompression is seen as a better alternative
* Heart or lung disease
* Any kind of systematic or local disease or illness that may significantly increase the risk of complications for the procedure related to injection
* Psychiatric illness that hinders participation in the study
* Known pregnancy or breast feeding
* Inadequate use of contraceptives
* Overuse or abuse of opioids
* Abuse of medications, narcotics or alcohol
* Anomalies which hinder or impede the used method of injection
* Allergy or any other hypersensitivity reactions against marcain, lidocaine, xylocain or adrenalin, botulinum toxin type A, Botox or any of it's constituents or any other related medication
* Treatment with medication that can interact with botulinum toxin type A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | for the follow-up period of 12 weeks
  Number of adverse events. Registration of any adverse events categorized by probable relationship to drug or the procedure. Data obtained from the headache diaries as well as open questions during consultations.

SECONDARY OUTCOMES:
Number of attacks with trigeminal neuralgia | 12 weeks
Intensity of the attacks | 12 weeks
  expressed as score on Visual analogue scale (VAS) for pain
Number of attacks with trigeminal neuralgia per 4 weeks per patient | 12 weeks
Number of doses of analgesics per 4 weeks per patient | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erling A Tronvik, PhD, MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Crespi J, Bratbak D, Dodick DW, Matharu M, Jamtoy KA, Tronvik E. Pilot Study of Injection of OnabotulinumtoxinA Toward the Sphenopalatine Ganglion for the Treatment of Classical Trigeminal Neuralgia. Headache. 2019 Sep;59(8):1229-1239. doi: 10.1111/head.13608. Epub 2019 Jul 25. PMID 31342515